CLINICAL TRIAL: NCT04421664
Title: Preemptive Therapy for SARS-Coronavirus-2 (COVID-19 PEP Canada)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Request of Health Canada after publication of https://doi.org/10.7326/M20-4207
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of Manitoba (Other); University of Alberta (Other); University of British Columbia (Other); McMaster University (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Eastern Health (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-6549
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Infection; SARS-CoV Infection; Coronavirus
Keywords: COVID-19; SARS-COV-2; Coronavirus; Corona virus
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Participants in this arm will receive the study drug, hydroxychloroquine.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo treatment.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — 200mg tablet; 800 mg orally once, followed in 6 to 8 hours by 600 mg, then 600mg once a day for 4 consecutive days
  Arms: Treatment
Drug: Placebo oral tablet — 4 placebo tablets once, followed in 6 to 8 hours by 3 tablets, then 3 tablets once-a-day for 4 consecutive days
  Arms: Placebo

SUMMARY:
Study Objective:

To test if early preemptive hydroxychloroquine therapy can prevent disease progression in persons with known symptomatic COVID-19 disease, decreasing hospitalizations and symptom severity.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a rapidly emerging viral infection causing COVID19. Therapy is generally not given to persons who are not hospitalized.

Hydroxychloroquine may have antiviral effects against SARS-CoV2 which may decrease disease severity when given early. This trial will use a modification of standard malaria dosing of hydroxychloroquine to provide preemptive therapy for those with early symptoms.

This study is a continuation of NCT04308668 which looked at post-exposure prophylaxis (now closed) and early treatment in the USA (now closed, data to be pooled) and Canada (which continues in this study). On April 28, 2020 NCT04308668 changed its primary outcome to symptomatic improvement in the preemptive therapy arm. This study continues enrollment for the primary ordinal outcome of hospitalization; hospitalization with intensive care stay; or death.

People in the participating Canadian provinces can help answer this critically important question. No in-person visits are needed.

The doses of hydroxychloroquine being used have been approved by Health Canada.

This trial is targeting the following groups of people:

If you are symptomatic with a positive COVID-19 test within the first 4 days of symptoms and are not hospitalized; OR If you have had occupational exposure with known exposure to someone with lab-confirmed COVID-19 within the last 14 days AND have compatible symptoms starting within the last 4 days;

You may participate if you live anywhere in the Canadian Provinces of Quebec, Manitoba, Alberta, British Columbia, Newfoundland or Ontario.

For information on how to participate in the research trial, go to:

www.covid-19research.ca

ELIGIBILITY:
Inclusion Criteria:

Age 18 years of age or older AND provision of informed consent

WITH

Symptomatic COVID-19 disease with confirmed diagnosis with PCR+ SARS-CoV-2 within <= 4 days of symptoms

OR

Healthcare worker with compatible symptoms with exposure to known PCR+ case <= 14 days (and no available/pending testing for the individual).

Exclusion Criteria:

* Current hospitalization
* Allergy to chloroquine or hydroxychloroquine
* Severe diarrhea and/or vomiting
* Significant hepatic impairment defined as known cirrhosis with history of hepatic encephalopathy or ascites.
* Prior retinal eye disease
* Concurrent malignancy requiring chemotherapy
* Known Chronic Kidney disease, Stage 4 or 5 or dialysis.
* Known glucose-6 phosphate dehydrogenase (G6PD) deficiency.
* Known ventricular arrythmia, known prolonged QTc interval, or any known episode of sudden cardiac death
* Known Porphyria
* Weight <40 kg
* Known Pregnancy of Breastfeeding
* Current use of chloroquine or hydroxychloroquine
* Current use of Artemether, Dapsone, Lumefantrine or Mefloquine
* Current use of Cardiac medicines: amiodarone, digoxin, dofetilide, flecainide, procainamide, sotalol, or propafenone
* Current use of the following antimicrobials: levofloxacin, ciprofloxacin, moxifloxacin, azithromycin, clarithromycin, erythromycin, ketoconazole, or itraconazole
* Current use of the following antidepressants: amitriptyline, citalopram, desipramine, escitalopram, imipramine, doxepin, fluoxetine, sertraline, bupropion (Wellbutrin), or venlafaxine
* Current use of the following antipsychotic or mood stabilizers: haloperidol, droperidol, lithium, quetiapine, thioridazine, ziprasidone
* Current use of methadone
* Current use of Sumatriptan, Zolmitriptan other than "as needed"
* Current use of systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Ordinal Scale of COVID19 Disease Severity at 14 days | 14 days
  Participants will self-report disease severity status as one of the following 3 options; no COVID19 illness (score of 1), COVID19 illness with no hospitalization (score of 2), or COVID19 illness with hospitalization or death (score of 3). Increased scale score indicates greater disease severity. Outcome is reported as the percent of participants who fall into each category per arm.

SECONDARY OUTCOMES:
Incidence of Hospitalization | 14 days
  Outcome reported as the number of participants in each arm who require hospitalization for COVID19-related disease.
Incidence of COVID-19 related Death | 90 days
  Outcome reported as the number of participants in each arm who expire due to COVID-19-related disease.
Incidence of all-cause Death | 90 days
  Outcome reported as the number of participants in each arm who expire due to all causes.
Incidence of All-Cause Study Medicine Discontinuation or Withdrawal | 14 days
  Outcome reported as the number of participants in each arm who discontinue or withdraw medication use for any reason.
Overall symptom severity at 5 and 14 days | 5 and 14 days
  Visual Analog Scale 0-10 score of rating overall symptom severity (0 = no symptoms; 10 = most severe)
Overall change in disease severity over 14 days among those who are symptomatic at baseline | 14 days
  Repeated Measure mixed regression model of change in: Visual Analog Scale 0-10 score of rating overall symptom severity (0 = no symptoms; 10 = most severe)

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD MPH FIDSA, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (8):
- University of Minnesota, Minneapolis, Minnesota, United States
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Eastern Health, St. John's, Newfoundland and Labrador
  - McMaster University, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset will be included with publication.
Supporting Information: Study Protocol, SAP
Time Frame: At time of publication
Access Criteria: To be publicly provided

REFERENCES:
- [Background] Skipper CP, Pastick KA, Engen NW, Bangdiwala AS, Abassi M, Lofgren SM, Williams DA, Okafor EC, Pullen MF, Nicol MR, Nascene AA, Hullsiek KH, Cheng MP, Luke D, Lother SA, MacKenzie LJ, Drobot G, Kelly LE, Schwartz IS, Zarychanski R, McDonald EG, Lee TC, Rajasingham R, Boulware DR. Hydroxychloroquine in Nonhospitalized Adults With Early COVID-19 : A Randomized Trial. Ann Intern Med. 2020 Oct 20;173(8):623-631. doi: 10.7326/M20-4207. Epub 2020 Jul 16. PMID 32673060
- [Background] Boulware DR, Pullen MF, Bangdiwala AS, Pastick KA, Lofgren SM, Okafor EC, Skipper CP, Nascene AA, Nicol MR, Abassi M, Engen NW, Cheng MP, LaBar D, Lother SA, MacKenzie LJ, Drobot G, Marten N, Zarychanski R, Kelly LE, Schwartz IS, McDonald EG, Rajasingham R, Lee TC, Hullsiek KH. A Randomized Trial of Hydroxychloroquine as Postexposure Prophylaxis for Covid-19. N Engl J Med. 2020 Aug 6;383(6):517-525. doi: 10.1056/NEJMoa2016638. Epub 2020 Jun 3. PMID 32492293
- [Background] Lother SA, Abassi M, Agostinis A, Bangdiwala AS, Cheng MP, Drobot G, Engen N, Hullsiek KH, Kelly LE, Lee TC, Lofgren SM, MacKenzie LJ, Marten N, McDonald EG, Okafor EC, Pastick KA, Pullen MF, Rajasingham R, Schwartz I, Skipper CP, Turgeon AF, Zarychanski R, Boulware DR. Post-exposure prophylaxis or pre-emptive therapy for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2): study protocol for a pragmatic randomized-controlled trial. Can J Anaesth. 2020 Sep;67(9):1201-1211. doi: 10.1007/s12630-020-01684-7. Epub 2020 May 7. PMID 32383125